CLINICAL TRIAL: NCT04997824
Title: Artificial Intelligence Guided Patient Selection for Atrial Fibrillation Catheter Ablation: Randomized Clinical Trial (AI-PAFA Trial)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2021-0608
Record Dates: First submitted 2021-07-19; First posted 2021-08-10 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Nutrition Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artificial Intelligence-based atrial fibrillation catheter ablation (Experimental): catheter ablation
  Interventions: Procedure: Artificial Intelligence-based atrial fibrillation catheter ablation
- Medical Therapy (Active Comparator): catheter ablation
  Interventions: Procedure: Medical Therapy

INTERVENTIONS:
Procedure: Artificial Intelligence-based atrial fibrillation catheter ablation — 1. Patient selection for Atrial Fibrillation Catheter Ablation(AFCA)
  2. AI-guided prediction for poor responder of AFCA in the outpatient clinic
  3. Sharing information on the AI prediction with the patient and family member
  4. AFCA after consent to the procedure
  5. Pulmonary vein isolation and additional treatment for non-pulmonary vein triggers
  6. Monitoring esophageal temperature
  7. Evaluation of Procedure and ablation time, and complication afer procedure
  8. Post-procedure rhythm follow-up is carried out according to the study design above.
  Arms: Artificial Intelligence-based atrial fibrillation catheter ablation
Procedure: Medical Therapy — 1. Patient selection for Atrial Fibrillation Catheter Ablation(AFCA)
  2. Decision for AFCA based on clinical guidelines and the experience of the attending physician
  3. AFCA after consent to the procedure
  4. Pulmonary vein isolation and additional treatment for non-pulmonary vein triggers
  5. Monitoring esophageal temperature
  6. Evaluation of Procedure and ablation time, and complication afer procedure
  Arms: Medical Therapy

SUMMARY:
Atrial fibrillation (AF) is a major cardiovascular disease with a prevalence of 1.7% of the total population in Korea, associated with 25% of ischemic stroke and 30% of heart failure, and is a major cardiovascular disease that doubles the risk of dementia. AF catheter ablation (AFCA) is an effective procedure that lowers the risk of heart failure mortality and cerebral infarction and improves cognitive or renal functions. However, the recurrence rate after the procedure is relatively high, especially in patients with long-standing persistent AF in which atrial remodeling has already progressed. Research on the prediction of treatment efficacy using artificial intelligence (AI) is being actively conducted around the world. We predicted the AFCA poor responders who will progress to permanent AF despite AFCA among a total of 3,372 patients included in the Yonsei AF Ablation cohort and the 2nd independent cohort with a long-term follow-up through AI with area under curve (AUC) 0.943. Therefore, in this prospective randomized clinical study, the difference between the patient selection for AFCA using AI algorithm and the clinical guidelines-based decision will be compared and evaluated in terms of long-term rhythm outcome.

DETAILED DESCRIPTION:
Study design

1. Prospective randomization (AI-based patient selection group vs. conventional guidelines-based patient selection group)
2. Target number of subjects 1000 patients (500 people in each group)
3. Rhythm follow-up schedule: 2012 ACC/AHA/ESC guidelines (basal, 3 months, then every 6 months Holter, ECG when symptomatic)
4. Anticoagulant therapy follows 2020 ESC guidelines.
5. Evaluation of all adverse events occurring in each group and comparative evaluation of hospitalization rates, major cardiovascular attacks, and mortality

Process of Patient Selection A guideline-based appropriate candidate for AFCA Randomization for AI-guide group vs. Clinical guideline-based group Poor responder selection by AI at the outpatient clinic AI-prediction outcomes should be noticed in AI-guided groups, but not in the clinical guideline-based group.

Recommendation of rate control for AI-predicted poor responders All-comer ablation in guideline-based group

Progress and rhythm/ECG tracking

1. Implemented according to 2012 American College of Cardiology(ACC)/American Heart Association(AHA)/Heart Rhythm Society(HRS) guidelines for AF management
2. Outpatient follow-up 1 to 2 weeks after the start of the procedure or drug treatment
3. Follow-up every 3 months after the procedure, and every 6 months thereafter
4. If the patient complains of arrhythmia symptoms, conduct an electrocardiogram at any time and follow the rhythm with a Holter or an event recorder.

ELIGIBILITY:
Inclusion Criteria:

1. Left atrium size < 55 mm
2. AF recurred during the administration of antiarrhythmic drugs or that antiarrhythmic drugs intolerable patients
3. Patients eligible for anticoagulant therapy (to prevent thromboembolic events)

Exclusion Criteria:

1. AF associated with severe cardiac anomalies or structural heart disease with hemodynamic influence
2. Patients who have difficulty in CT imaging using a contrast medium
3. Patients with active internal bleeding
4. Inappropriate anticoagulant therapy
5. Serious comorbidities
6. Patients expected to survive less than 1 year
7. People with drug or alcohol addiction
8. Those who cannot read the consent form (illiterate, foreigners, etc.)
9. Patients who are judged unsuitable for participation in clinical research by the judgment of other investigators

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-10-07 (Actual); Primary Completion 2031-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Atrial Fibrillation Catheter Ablation(AFCA) | Up to 5 years
  Efficacy evaluation: Clinical recurrence rate - Defined as AF or atrial tachycardia lasting over 30 seconds after 3 months of procedure. Rhythm monitoring based on 2012 ACC/AHA/HRS guidelines as described above. 24-hour Holter ECG monitoring will be performed at 2-3 month and every 6 months within 2 years of procedure, Holter every 1 year after 2 years of procedure and ECG and monitoring with a Holter or an event recorder will be performed at any time if the patient complains of symptoms
safety of Atrial Fibrillation Catheter Ablation(AFCA) | Up to 5 years
  Safety Assessment: Incidence of procedure-related complications within 30 days of procedure (thoracotomy, cerebral infarction, pericardial effusion or pericardial tamponade, inguinal puncture site hematoma, and vascular complications)

SECONDARY OUTCOMES:
Comparison of procedure time, ablation time and hospitalization period | Immediate after procedure
Anti-arrhythmic drug or anticoagulation therapy related complication rate | 1 week, 3, 6, 12, 18, 24, 36 months after procedure
Re-hospitalization rate of electrical cardioverson after the procedure | 1 week, 3, 6, 12, 18, 24, 36 months after procedure
number of electrical cardioversion after the procedure | 1 week, 3, 6, 12, 18, 24, 36 months after procedure
Major cardiovascular event rate - Death, myocardial infarction, coronary angioplasty, and re-hospitalization for arrhythmia and heart failure | Immediate after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Nam Pak, Principal Investigator — Severance Hospital, Yonsei University Health System
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided